CLINICAL TRIAL: NCT04604925
Title: A Pilot Study of Hypertension Management Using Remote Patient Monitoring
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Omron Healthcare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Professor of Medicine, Division of General Internal Medicine & Geriatrics, Northwestern University
Other Study IDs: STU00213093
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Remote Patient Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Remote patient monitoring for hypertension: RPM Integration: All intervention practices will receive communication by email explaining RPM procedures, ordering, use, and financial implications. We will also present this information at practice meetings. Primary care clinicians at these sites will receive clinical decision support (Epic Best Practice Alert) for patients meeting primary or secondary eligibility criteria. It will be at the discretion of the primary care clinicians when to offer or refer patients to RPM.
  Interventions: Behavioral: Remote patient monitoring for hypertension
- Usual care: Matching patients from control practices will be selected from remaining Northwestern Medical Group primary care sites and be chosen to provide as sufficiently large number of eligible patients for comparison. These groups will contribute EHR data through the NM EDW but will not have any new procedures put in place

INTERVENTIONS:
Behavioral: Remote patient monitoring for hypertension — Intervention involves practices making available remote physiologic monitoring treatment management services allowable under Medicare for blood pressure (and weight if desired) to Medicare patients in the practice when ordered by the patient's clinician.
  Groups: Remote patient monitoring for hypertension

SUMMARY:
The investigators will conduct a pragmatic pilot test of a remote patient monitoring system (RPM) for blood pressure measurement for Medicare patients with hypertension. The primary objective is to better understand how patients' remote monitoring of blood pressure and the direct transmission of this data to a healthcare system's EHR can be used by the patient and the care team to support optimal hypertension care.

This pilot study which we will conduct in two Northwestern Medical Group (NMG) primary care practices will: evaluate the integration of Omron's remote monitoring system into Northwestern Medicine's electronic health record (so that clinical data can flow directly from the patient's monitor to the EHR), evaluate the use of billing work flows for covered Medicare services, build and deploy clinical decision support to aid with patient identification and ordering of the remote patient monitoring system, and evaluate the uptake and clinical effects of this system in the pilot practices compared to matched patients selected from non-pilot control practices.

The investigators will conduct a pragmatic non-blinded, non-randomized pilot study with contemporaneous controls among NMG outpatient clinics that provide adult primary care. They will make comparisons of data obtained through the course of routine care delivery from pilot and non-pilot practices.

DETAILED DESCRIPTION:
Investigators at Northwestern University will partner with Omron Healthcare Co., Ltd. (hereinafter referred to as "Omron") to conduct a pragmatic pilot test of a remote patient monitoring system (RPM) for blood pressure measurement for Medicare patients with hypertension. The primary objective is to better understand how patients' remote monitoring of blood pressure and the direct transmission of this data to a healthcare system's EHR can be used by the patient and the care team to support optimal hypertension care. The procedures that will be evaluated are routine healthcare services that are currently reimbursable by Medicare. However, the optimal ways to: integrate these tools into primary care practice, promote clinician and patient uptake, and put this information to use in the clinical environment to best control hypertension are not fully understood. This pilot study which we will conduct in two Northwestern Medical Group (NMG) primary care practices will: evaluate the integration of Omron's remote monitoring system into Northwestern Medicine's electronic health record (so that clinical data can flow directly from the patient's monitor to the EHR), evaluate the use of billing work flows for covered Medicare services, build and deploy clinical decision support to aid with patient identification and ordering of the remote patient monitoring system, and evaluate the uptake and clinical effects of this system in the pilot practices compared to matched patients selected from non-pilot control practices.

The remote patient monitoring (RPM) system will be provided by Omron Healthcare to eligible patients at no charge. This will include a Bluetooth enabled home blood pressure monitor, a simplified smart phone connected to the Verizon network and, if requested, a Bluetooth enabled scale. Patients who are agreeable to using this RPM system will have this service ordered by their clinician will have this equipment mailed to their homes. Payments for reimbursable remote monitoring services will be billed by Northwestern Medicine to Medicare and supplemental insurance coverage in the fashion that is permitted under Medicare rules.

The investigators will conduct a pragmatic non-blinded, non-randomized pilot study with contemporaneous controls among NMG outpatient clinics that provide adult primary care. We will make comparisons of data obtained through the course of routine care delivery from pilot and non-pilot practices.

ELIGIBILITY:
Inclusion Criteria:We will use these criteria to determine which patients will be included or excluded in the study analytic data set.

General inclusion criteria:

* Adults aged 65 to 85 years at the time of the study start date
* Receive their primary care from an eligible Northwestern Medicine clinic site
* One or more office or telehealth visits in the year preceding the study start date

Inclusion criteria primary population:

* Last two office blood pressures ≥140 mm Hg systolic or ≥90 mmHg diastolic
* Diagnosis of hypertension in the year preceding the study start date (problem list or encounter diagnosis)

Inclusion criteria for secondary population

* Meet criteria for primary population OR
* Diagnosed hypertension but did not have the last two office blood pressures ≥140 mm Hg systolic or ≥90 mmHg diastolic OR
* No diagnosis of hypertension in the past year but did have the last office blood pressure ≥140 mm Hg systolic or ≥90 mmHg diastolic

Exclusion Criteria: • Persistent atrial fibrillation as indicated in the electronic health record (EHR)

* Stage IV or more severe kidney disease, defined as estimated glomerular filtration rate <30 per 1.73 m2 or currently on renal replacement therapy (i.e. hemodialysis or peritoneal dialysis)
* Diagnosis of dementia as indicated in the electronic health record

Ages: 65 Years to 85 Years | Sex: All
Age Groups: Older Adult
Study Population: This study will take place in several Northwestern Medicine Group outpatient primary care clinic settings. Patients at these practices will be eligible for inclusion in the primary study population if they have diagnosed hypertension, are 65 to 85 years old, have Medicare insurance, and have their last two prior office blood pressures ≥140 mm Hg systolic or ≥90 mm Hg diastolic. Patients at these practices will be eligible for inclusion in the secondary study population if either they meet the inclusion criteria for the primary population or they are 65 to 85 years old, have Medicare insurance and either have diagnosed hypertension but do not have their last two office blood pressures prior ≥140 mm Hg systolic or ≥90 mm Hg diastolic, or they do not have hypertension diagnosed and have their most recent prior office blood pressure ≥140 mm Hg systolic or ≥90 mm Hg diastolic.
Sampling Method: Non-Probability Sample
Enrollment: 7068 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Performance measure Controlling High Blood Pressure (NQF 0018) | 6 months
  Proportion of eligible hypertension patients with most recent eligible blood pressure in the measurement period <140/90 mm Hg
Systolic blood pressure at the most recent office visit | 6 months
  Systolic blood pressure at the most recent office visit (mm Hg)

SECONDARY OUTCOMES:
Antihypertensive medication intensification | 6 months
  Antihypertensive medication intensification
Antihypertensive medication intensification | 3 months
  Antihypertensive medication intensification
Performance measure Controlling High Blood Pressure (NQF 0018) | 3 month
  Proportion of eligible hypertension patients with most recent eligible blood pressure in the measurement period <140/90 mm Hg
Performance measure Controlling High Blood Pressure (NQF 0018) | 1 month
  Proportion of eligible hypertension patients with most recent eligible blood pressure in the measurement period <140/90 mm Hg
Systolic blood pressure at the most recent office visit | 3 months
  Systolic blood pressure at the most recent office visit (mm Hg)
Systolic blood pressure at the most recent office visit | 1 month
  Systolic blood pressure at the most recent office visit (mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Persell, MD/MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Division of General Internal Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Petito LC, Anthony L, Peprah YA, Lee JY, Li J, Sato H, Persell SD. Remote physiologic monitoring for hypertension in primary care: a prospective pragmatic pilot study in electronic health records using propensity score matching. JAMIA Open. 2023 Jan 31;6(1):ooac111. doi: 10.1093/jamiaopen/ooac111. eCollection 2023 Apr. PMID 36743315

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT04604925/SAP_000.pdf